CLINICAL TRIAL: NCT05773352
Title: Tornier Perform® Humeral System - Fracture Study
Brief Title: Perform® Humeral System - Fracture Study (PFX)
Acronym: PFX
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: UE-01-2022
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Arthropathy of Shoulder; Fracture Humerus; Traumatic Arthritis; Revision of Other Devices if Sufficient Bone Stock Remains
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Tornier Perform® Humeral System - Fracture: Commercially available convertible humeral system for anatomic and reverse shoulder arthroplasty.
  Interventions: Device: Tornier Perform® Humeral System - Fracture

INTERVENTIONS:
Device: Tornier Perform® Humeral System - Fracture — A replacement of shoulder joints for anatomic and reverse shoulder arthroplasty.
  A replacement of other shoulder joints devices in case of revisions if sufficient bone stock remains.

SUMMARY:
This study is an international, single arm, multicenter, prospective follow-up, non-significant risk, Post-Market Clinical Follow-up (PMCF), which is designed to collect safety and performance data on commercially available Perform® Fracture.

Data collected from this study will be used for purposes, including but not limited to, PMS, peer-reviewed publications, education materials, future regulatory submissions, and/or product development.

DETAILED DESCRIPTION:
This is an International, single arm, multicenter, prospective follow-up, non-significant risk, Post-Market Clinical Follow-up (PMCF) study. Data will be collected for the commercially available Perform® Fracture shoulder system in both the anatomic and reversed configurations.

The primary endpoint of this study is to demonstrate decreased pain and improved subjects' shoulder functionality of daily living by achieving a mean of American Shoulder and Elbow Surgeons (ASES) shoulder score higher than 62 points, at 2-year follow-up post-operatively, regardless of configuration (anatomic or reverse).

Retrospective inclusions are allowed: preoperative, intra operative, and 6 months data can be collected retrospectively up to 12 months after the surgery date.

Secondary outcome measures include patient reported outcome measures (PROMs) and standard radiographic findings, including, but not limited to: bone erosion, device migration/subsidence, component breakage, radiolucency, and ossification.

Safety and performance data will be collected at surgery, immediate post-op, and up to 10 years post-operation. Patient Reported Outcome Measures (PROMs), device revision and Adverse Events (AEs) will be assessed annually throughout the study.

Range of Motion (ROM), strength and radiographic imaging assessments of the study shoulder will also be performed for in-person milestones visits at 6 months (radiographic imaging assessments), 1-, 2-, 5- and 10-year, post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of the informed consent or the non-opposition (when applicable)
* Informed and willing to sign an informed consent form (ICF) approved by IRB or EC (when applicable)
* Willing and able to comply with the requirements of the study protocol
* Considered a candidate for shoulder arthroplasty with the device for shoulder joint disabled by:

  * Traumatic or pathologic conditions of the shoulder resulting in fracture of the glenohumeral joint, including humeral head fracture and displaced 3-or 4-part proximal humeral fractures
  * Fracture sequelae
  * Revisions where adequate fixation can be achieved, and adequate bone stock remains after final reconstruction
  * Proximal humerus bone defect (reverse configuration)

Exclusion Criteria:

* Not able to comply with the study procedures based on the judgment of the assessor (e.g., cannot comprehend study questions, inability to keep scheduled assessment times)
* Patient belongs to a vulnerable group of subjects, including minor subjects, those unable to decide for themselves to participate or needing a LAR, or others who could be subject to coercion (subjects who may not be acting on their own initiative) (referred as "vulnerable subject" in the section 3.44 of the ISO 14155:2011 norm)
* Any absolute contraindications as mentioned in the device Instruction For Use (available on ifu.stryker.com)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 120 subjects are to be enrolled in this clinical investigation. Subjects participating in this clinical investigation will be recruited from the investigator's standard subject population, where all subjects presenting for an anatomic or reverse shoulder arthroplasty will be evaluated for clinical investigation participation based on the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
ASES Score = American Shoulder and Elbow Surgeons Score | 24 Month
  11 items with total score reported out of 100 measuring pain and activity of patient's evaluated shoulder where lower scores indicate more pain and less function

SECONDARY OUTCOMES:
Constant Score | 24 Month
  A score based on a 100-point scale determined by objective measurements made by the physician in the clinic and subjective values based on pain and activities of daily living reported by the patient. Collected at: 1, 2, 5, and 10 years.
SANE | 24 Month
  Single question that asks the patient to rate their shoulder on a scale from 0 to 100, where 100 is normal. Collected annually through 10 year visit.
EQ-5D-5L | 24 Month
  Consists of a 5-question measure where patients rate their health today on a 5-point scale on a 5-dimension scale and a visual analogue scale to measure overall health status. Collected annually through 10 year visit..
Patient Satisfaction | 24 Month
  Single subjective question "How satisfied are you with your shoulder?" Collected annually through 10 year visit.
Radiographic Findings | 24 Month
  X-rays will be analyzed, when sufficient information is available, for bone erosion, device migration/subsidence, component breakage, radiolucency, and ossification. X-rays will be collected at Baseline, 6 months, 1 year, 2 year, 5 year and 10 year.
Tuberosity healing | 12 Month
  Tuberosity healing (bone union) (Boileau et al., 2002, 2013, 2019) is expected to be completed post-operatively at 6 months and assessed at 6 months and up to 1 year if tuberosity healing is not achieved at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (9):
- United States (9):
  - More Foundation, Phoenix, Arizona
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Eisenhower Health Desert Orthopedic Center, Rancho Mirage, California
  - California Pacific Orthopaedics, San Francisco, California
  - The Center for Bone and Joint Disease, Hudson, Florida
  - Loyola University Chicago, Maywood, Illinois
  - Washington University, St Louis, Missouri
  - Tennessee Orthopaedic Alliance, Columbia, Tennessee
  - University of Texas/UT Health, Houston, Texas

IPD SHARING:
Plan to Share IPD: No